CLINICAL TRIAL: NCT00000600
Title: Antioxidants and Prevention of Early Atherosclerosis
Brief Title: Vitamin E and C to Slow Progression of Common Carotid Artery Plaque Build-Up
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 106; U01HL052073 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2006-10

CONDITIONS: Cardiovascular Diseases; Carotid Artery Diseases; Intracranial Arteriosclerosis; Cerebrovascular Disorders; Heart Diseases; Vascular Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Carotid Artery Diseases; Intracranial Arteriosclerosis; Cerebrovascular Disorders; Heart Diseases; Vascular Diseases; Atherosclerosis | interventions — Vitamin E; Ascorbic Acid

INTERVENTIONS:
Drug: Vitamin E
Drug: Vitamin C

SUMMARY:
This study will evaluate the effects of vitamin E supplementation in retarding the progression of common carotid artery intima-media thickening in African Americans.

DETAILED DESCRIPTION:
BACKGROUND:

Evidence from epidemiologic studies, and from one unpublished study, suggests that greater intake of antioxidant vitamins is associated with reduced risk of coronary heart disease and stroke. Findings from an animal model indicate that increased intake of antioxidant vitamins prevents progression of aortic fatty streaks induced by an atherogenic diet, but not from more advanced injury-induced lesions. These observations suggest the hypothesis that increased antioxidant vitamin intake may prevent further progression of early atherosclerosis, possibly by means of reduced susceptibility of low density lipoprotein to oxidative modification and consequent cytotoxic, chemotactic, chemostatic, and unregulated uptake effects.

A new, automated, low-cost, portable ultrasound system for determining intima-media thickness of the common carotid artery makes it feasible to test the primary prevention impact of antioxidant vitamins on early atherosclerosis. Results of two studies at the University of Southern California suggest that the low-density lipoprotein effects on common carotid artery intima-media thickness can be detected by automated methods within 12 to 24 months in small patient samples. Retardation of intima-media thickness progression was achieved in both studies without significant changes in average vessel diameter, which suggests effects on early atherosclerotic lesions.

DESIGN NARRATIVE:

Patients will be screened for carotid intima-media thickness at home or at schools in mobile vans equipped with portable ultrasound equipment. After 12 months, those patients above the age and sex-adjusted 66th percentile at Screen I will be re-screened (Screen II), and those showing the greatest progression in intima-media thickness will be invited to participate in a trial run-in to assess vitamin E compliance. Patients will be randomized to the following four groups: 1) vitamin E (573 mg/day); 2) vitamin C; 3) Vitamin E and C combined; and 4) placebo. Common carotid artery intima-media thickness will be observed by ultrasound at 12- and 24-month follow-ups. The primary outcome is 24-month rate of change in average common carotid artery intima-media thickness.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Inclusion Criteria:

* African American

Ages: 35 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1995-06; Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
rate of change in average common carotid artery intima-media thickness (measured over 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: James H. Dwyer, III, Principal Investigator — University of Southern California